CLINICAL TRIAL: NCT04848324
Title: Short-Term Effectiveness of Ultrasound-Guided Corticosteroid Hydrodissection in Patients With Carpal Tunnel Syndrome
Brief Title: Short-Term Effectiveness of Ultrasound-Guided Corticosteroid Hydrodissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; ultrasonography; hydrodissection; steroid injection
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): 14 patients (14 hands) who received US-guided corticosteroid hydrodissection
  Interventions: Other: Corticosteroid Hydrodissection
- Control group (Active Comparator): 14 patients (14 hands) who received US-guided corticosteroid injection
  Interventions: Other: Corticosteroid Injection

INTERVENTIONS:
Other: Corticosteroid Hydrodissection — The median nerve was examined by US at the scaphoid-pisiform level of the inlet of carpal tunnel. The hydrodissection was achieved by a total volume of 3 mL (1 mL of triamcinolone and 2 mL of saline) in the intervention group based on a study identifying median nerve hydrodissection with this volume. Half of the total volume (1.5 mL ) was delivered via the in-plane ulnar approach and the other half (1.5 mL) via the in-plane median approach to create a fluid plane along the nerve.
  Arms: Intervention group
Other: Corticosteroid Injection — 1 mL of triamcinolone was delivered via the in-plane ulnar approach
  Arms: Control group

SUMMARY:
Aim: Steroid injections are remarkably effective as a treatment for carpal tunnel syndrome (CTS) in the short term. The aim of this study was to determine whether hydrodissection would provide an additional clinical effect when used along with a corticosteroid in the short term.

Methods: A prospective cohort of patients with CTS were retrospectively evaluated. 28 patients were selected randomly who received ultrasound (US)-guided triamcinolone hydrodissection (3 mL) as intervention group and received US-guided triamcinolone injection (1 mL) as control group, from the data (case-control ratio 1:1). Outcome measures were the Boston Carpal Tunnel Questionnaire (BCTQ), hand grip strength (HGS), fhe cross-sectional area (CSA) of the median nerve and Short Form 12 (SF-12). Assessments were recorded at baseline, 1 and 4 weeks after injection.

DETAILED DESCRIPTION:
Background: Steroid injections are remarkably effective as a treatment for carpal tunnel syndrome (CTS) in the short term.

Aim: To determine whether hydrodissection would provide an additional clinical effect when used along with a corticosteroid in the short term.

Methods: A prospective cohort of patients with CTS were retrospectively evaluated. 28 patients were selected randomly who received ultrasound (US)-guided triamcinolone hydrodissection (3 mL) as intervention group and received US-guided triamcinolone injection (1 mL) as control group, from the data (case-control ratio 1:1). Outcome measures were the Boston Carpal Tunnel Questionnaire (BCTQ), hand grip strength (HGS), fhe cross-sectional area (CSA) of the median nerve and Short Form 12 (SF-12). Assessments were recorded at baseline, 1 and 4 weeks after injection.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18-65
2. clinically diagnosed with CTS
3. electrophysiologically confirmed mild-to-moderate CTS
4. having typical CTS symptoms for at least 3 months
5. not benefiting from splinting and resting.

Exclusion Criteria:

1. electrophysiologically diagnosed with severe CTS
2. surgery history for CTS
3. presence of metabolic, endocrine and neoplastic disorders
4. presence of other neurological disorders (such as plexopathy, cervical radiculopathy, proximal median or ulnar neuropathy, polyneuropathy and mononeuritis multiplex)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | baseline, change from baseline BCTQ at 1 and 4 weeks after injection
  The Boston Carpal Tunnel Questionnaire (BCTQ) consisting of two subscales (Symptom Severity Scale (SSS) and Functional Status Scale (FSS)) was filled out by the patient him/herself. Both subscales of BCTQ are scored between 1 and 5, and higher scores illustrate a greater degree of disability. The Turkish validity of the questionnaire was demonstrated.
Hand grip strength (HGS) | baseline, change from baseline HGS at 1 and 4 weeks after injection
  The Standard Jamar Dynamometer was used to measure HGS. The patients were placed in a sitting position with the forearm in a neutral position and the elbow in 90 ° flexion. Three consecutive measurements were performed and the average value of the measurements were noted. Studies have shown that the Jamar dynamometer has high validity and reliability and is considered to be the gold standard for evaluating HGS
Cross-Sectional Area of the Median Nerve | baseline, change from baseline CSA at 1 and 4 weeks after injection
  The cross-sectional area (CSA) of the median nerve was measured at the scaphoid-pisiform level by using US since the swelling of the median nerve is a reliable measure for post-injection follow-up at this level (Figure 3). Three measurements were done and averaged for analysis.

SECONDARY OUTCOMES:
Short Form 12 (SF-12) | baseline, change from baseline SF-12 at 1 and 4 weeks after injection
  Quality of life was assessed with the Turkish version of Short Form 12 (SF-12). A physical component score and a mental component score are obtained from the SF-12. Higher scores show better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Orucu Atar, Principal Investigator — Gaziler Physical Medicine and Rehabilitation, Training and Research Hospital, Department of PMR
Locations (1):
- Merve Orucu Atar, Ankara, Cankaya, Turkey (Türkiye)